CLINICAL TRIAL: NCT03828513
Title: Can the Effects of High Flow Nasal Cannula Oxygenation on Postoperative Atelectasis be Evaluated With Lung Ultrasound: A Randomized Controlled Prospective Study
Brief Title: Can the Effects of High Flow Nasal Cannula Oxygenation on Postoperative Atelectasis be Evaluated With Lung Ultrasound
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, EMİNE YURT, Principal Investigator, Kocaeli Derince Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: KIA 2018/174
Record Dates: First submitted 2018-12-22; First posted 2019-02-04 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Atelectasis; Bariatric Surgery Candidate; Ultrasound Therapy; Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow nasal cannula oxygen applied (Active Comparator): High flow nasal cannula oxygen is start at a flow rate of 80 L/min with 100% oxygen in the preoperative period.
  Interventions: Device: High flow nasal cannula oxygen is applied
- High flow nasal cannula oxygen is not applied (Active Comparator): Preoxygenation will be applied with an oxygen supplement of 5 l/min to an endtidal O2> 90%.
  Interventions: Device: High flow nasal cannula oxygen is not applied

INTERVENTIONS:
Device: High flow nasal cannula oxygen is applied — Atelectasis evaluation with lung ultrasound is performe and score in 6 different areas before and after High flow nasal cannula oxygen. Pulmonary function tests and blood gas parameters are compared.During the procedure, the patient's blood pressure, heart rate, oxygen saturation, any complications that may develop will be recorded.Induction of anesthesia; difficult airway management, difficult mask and / or difficult intubation incidence, Mallampati scores, the use of one of the difficult intubation techniques during intubation, perioperative mechanical ventilation parameters (ventilation mode, tidal volume, respiratory frequency, end of tidal CO2 (carbon dioxide) pressure, PEEP usage, SpO2 (saturation oxygen), airway peak pressure, urine volume, arterial blood gas parameters are recorded.
  Arms: High flow nasal cannula oxygen applied
Device: High flow nasal cannula oxygen is not applied — Apply preoxygenation with facemask. Prior to induction of general anesthesia, preoxygenation will be applied with an oxygen supplement of 5 l / min to an endtidal O2> 90%.Atelectasis evaluation with lung ultrasound is performe and score in 6 different areas before and after preoxygenation.
  Arms: High flow nasal cannula oxygen is not applied

SUMMARY:
Evaluate the effects of high-flow nasal oxygen therapy on atelectasis in the perioperative period by lung ultrasound (LUS) in bariatric surgery patients.

DETAILED DESCRIPTION:
In obese patients, lung compliance decreases by 25% and Functional Residual Capacity decreases by about one-third. As they consume about 25% more oxygen than non-obese individuals, postoperative pulmonary complications occur more commonly. POINT (Peri-Operative Insufflatory Nasal Therapy) provides humidified and heated high flow oxygen therapy in perioperative period. High-ﬂow nasal oxygen (HFNO) facilitates oxygenation and ventilation of both the spontaneously breathing and apnoeic patient.High-ﬂow nasal cannula oxygen came to prominence in anaesthesia when it was shown to prolong the time to oxygen desaturation in patients with a difﬁcult airway.

Lung ultrasonography (LUS) has been used more frequently in the diagnosis of pulmonary pathologies than chest radiography. This prospective observational study is to evaluate the effects of high-flow nasal oxygen therapy on atelectasis in the perioperative period by lung ultrasound (LUS) in bariatric surgery patients.

Materials and Methods: Following the Ethics Committee approval and written informe consents, 100 adult bariatric surgery patients are include in this observational study. The patients are randomly distributed into two groups ; High Flow Nasal Cannula Oxygenation(HFNCO) made group(n:50); HFNCO not made group(n:50).

HFNCO is start at a flow rate of 20 L/min with 100% oxygen in the preoperative period. It is titrate up to 50 L/min and increase to 80 L/min under general anesthesia until tracheal intubation. Atelectasis evaluation with lung ultrasound is performe and score in 6 different areas before and after HFNCO.

Pulmonary function tests and blood gas parameters are compared.During the procedure, the patient's blood pressure, heart rate, oxygen saturation, any complications that may develop will be recorded.nduction of anesthesia; difficult airway management, difficult mask and / or difficult intubation incidence, Mallampati scores, the use of one of the difficult intubation techniques during intubation (such as FastTrack, videolaryngoscopy or fiberoptic intubation), perioperative mechanical ventilation parameters (ventilation mode, tidal volume, respiratory frequency, end of tidal CO2 (carbon dioxide) pressure, PEEP usage, SpO2 (saturation oxygen), airway peak pressure, urine volume, arterial blood gas parameters are recorded.Duration of operation, surgical method (laparotomy / laparoscopy), agents used in induction and postoperative analgesia, use of blood, blood product and vasopressor are recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Above 18 years;
2. Patients who have undergone obesity surgery;
3. ASA 2-3 patients;
4. Patients who have received written informed consent;

Exclusion Criteria:

1. Patients under the age of 18;
2. Patients refusing to participate in the study;
3. Patients under emergency conditions;
4. Earlier laryngeal and tracheal surgery;
5. allergies to lidocaine;
6. Patients with FEV1 / FVC below 60%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 Years to 80 Years (Adult, Older Adult)
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of postoperative atelectasis in bariatric surgery patients | Up to 20 minutes in postoperative care unit
  Postoperative atelectasis develops in patients undergoing laparoscopic bariatric surgery under anesthesia.After the operation a researcher will perform lung ultrasonography postoperative at minute 5. reseracher will detect 6 region of each lung totally 12 regions. the researcher will record the modified and original lung ultrasonography scores (LUS score) of the patients. LUS Score is a scoring system to eveluate atelectasis of lung and scores 1-3 points for each region (min score 0 max score 36)

CONTACTS AND LOCATIONS:
Overall Officials: Emine Yurt, doctor, Principal Investigator — Investigator
Locations (1):
- Kocaeli Derince Education and Research Hospital, Kocaeli, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No